CLINICAL TRIAL: NCT05270005
Title: Progression Assessment of Carotid Artery Stenosis by Ultrafast Ultrasound Flow Imaging
Acronym: CAS-PRO
Status: Active, not recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1915
Record Dates: First submitted 2022-02-02; First posted 2022-03-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Carotid Artery Stenosis
Keywords: Ultrafast ultrasound flow imaging; Atherosclerotic plaque; Disease progression; Velocity vector imaging
MeSH Terms: conditions — Carotid Stenosis; Plaque, Atherosclerotic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic carotid artery stenosis: Patients with an asymptomatic carotid artery stenosis, defined by 30% to 69% narrowing of the carotid artery according to conventional duplex measurements in the absence of ipsilateral retinal or cerebral ischemia in the preceding 6 months.
  Interventions: Diagnostic Test: Ultrasound-based flow imaging; Diagnostic Test: Ultrasound-based strain imaging; Diagnostic Test: Conventional duplex

INTERVENTIONS:
Diagnostic Test: Ultrasound-based flow imaging — Ultrasound-based flow imaging of the carotid artery stenosis will be acquired at baseline and two annual follow-up appointments.
Diagnostic Test: Ultrasound-based strain imaging — Ultrasound-based strain imaging of the carotid artery stenosis will be acquired at baseline and two annual follow-up appointments.
Diagnostic Test: Conventional duplex — Conventional duplex measurements of the carotid artery stenosis will be acquired at baseline and two annual follow-up appointments.

SUMMARY:
Rationale: Approximately 15-20% of strokes originates from an atherosclerotic plaque rupture in the carotid artery. To reduce the risk of stroke, patients should be evaluated for possible carotid endarterectomy (CEA), which is based on simple geometrical and clinical measures. Multiple studies have shown that the current risk stratification may lead to both over- and under-treatment for patients with carotid artery stenosis. This implicates that the current guidelines are lacking patient-specific parameters and have limited sensitivity. There is a wealth of evidence implicating the important role of local (disturbed) blood flow throughout the onset and progression of atherosclerosis. Novel flow-related measures, that go beyond simple geometrical indications, are required to improve diagnosis and treatment in patients with carotid artery stenosis. Nowadays, ultrasound (US) is one of the main techniques to assess for the presence and extent of carotid artery stenosis. However, current clinically-used US systems are unable to acquire and visualize the complex flow phenomena that play such a crucial role in the atherosclerotic disease process. With the advent of ultrafast ultrasound imaging, acquiring thousands of images per second, continuous tracking of flow in all directions became feasible, which enables us to image two-dimensional blood flow and possible disturbances with high accuracy and precision.

In this project, we aim to assess whether flow (related) parameters are associated with disease progression (and if so, which), in order to map the progression of atherosclerotic plaques using non-invasive, US-based blood flow imaging. In the future, this could improve risk stratification for individual patients for surgery, decrease patient mortality and morbidity, and therefore reduce healthcare costs.

Objective: To longitudinally assess the association between spatio-temporal blood flow velocities (peak systole and end-diastole at common carotid artery, maximum stenosis and internal carotid artery) and the progression of carotid atherosclerosis defined by duplex measurements.

Secondary objectives are to investigate the association between blood flow-derived parameters, including wall shear stress (WSS), vector complexity and vorticity, and the progression of atherosclerosis defined by duplex measurements. Furthermore, to assess the association between spatio-temporal blood flow velocities and blood flow-derived parameters (WSS, vector complexity and vorticity) and the progression of atherosclerosis as measured using ultrasound-based strain imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (≥18 years old);
* Informed consent form understood and signed, and patient agrees to follow-up visits;
* Presence of carotid artery stenosis (between 30%-69%) according to conventional duplex measurements (peak-systolic velocity of 125-230 cm/s [5] in combination with visible lumen reduction >30% according to North American Symptomatic Carotid Endarterectomy Trial [NASCET] method);
* Defined asymptomatic with respect to the ipsilateral carotid artery stenosis.

Exclusion Criteria:

* A planned carotid revascularisation for the ipsilateral carotid artery stenosis at date of inclusion;
* History of carotid revascularisation at artery under investigation;
* Visible near occlusion at asymptomatic stenosis side according to conventional duplex measurements;
* Life expectancy < 2 years;
* Participating in another clinical study, interfering on outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an asymptomatic carotid artery stenosis, defined by 30% to 69% narrowing of the carotid artery according to conventional duplex measurements in the absence of ipsilateral retinal or cerebral ischemia in the preceding 6 months.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Two-dimensional spatio-temporal blood flow velocities | 2 year follow-up
  Two-dimensional vector velocity fields derived from the US-based flow imaging will be used to calculate the spatio-temporal blood flow velocities.
Plaque progression (stenosis degree) | 2 year follow-up
  Plaque progression, defined by increase in stenosis degree. Stenosis degree will be quantified by conventional ultrasound imaging.

SECONDARY OUTCOMES:
Wall shear stress | 2 year follow-up
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is the wall shear stress.
Vorticity | 2 year follow-up
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is vorticity.
Vector complexity | 2 year follow-up
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is vector complexity.
Plaque progression (deformation) | 2 year follow-up
  Plaque progression, defined by change in plaque deformation. Plaque deformation will be quantified by strain imaging.
Symptomatic carotid stenosis | 2 year follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - Radboud university medical center, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided